CLINICAL TRIAL: NCT05195268
Title: Reduction in Arrhythmia Burden With Left Atrial Posterior Wall Ablation for Persistent AF
Acronym: RABLAP-AF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision to discontinue in light of new evidence demonstrating that the intervention in question is not effective.
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Collaborators: Biosense Webster, Inc. (Industry); Royal Brompton & Harefield NHS Foundation Trust (Other); St George's University Hospitals NHS Foundation Trust (Other); University Hospital Plymouth NHS Trust (Other); South Tees Hospitals NHS Foundation Trust (Other); Manchester University NHS Foundation Trust (Other Government); Guy's and St Thomas' NHS Foundation Trust (Other); Papworth Hospital NHS Foundation Trust (Other Government); Portsmouth Hospitals NHS Trust (Other Government); University Hospitals Dorset NHS Foundation Trust (Other Government); University Hospital Birmingham NHS Foundation Trust (Other); Onze Lieve Vrouw Hospital (Other); AZ Sint-Jan AV (Other); University of Liverpool (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1349
Record Dates: First submitted 2021-11-19; First posted 2022-01-18 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Posterior wall isolation; Ablation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: A randomised controlled trial with two arms: 1) Pulmonary vein isolation + posterior wall isolation; 2) Pulmonary vein isolation alone
Who Masked: Outcomes Assessor
Masking Description: Patients and operators will be aware of the treatment arm. Researchers interpreting and assessing outcome data will be blinded to treatment received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - PVI + PWI (Active Comparator): These patients will receive pulmonary vein isolation and posterior wall isolation.
  Interventions: Procedure: Intracardiac Catheter Ablation
- Group 2 - PVI only (Other): These patients will receive pulmonary vein isolation only.
  Interventions: Procedure: Intracardiac Catheter Ablation

INTERVENTIONS:
Procedure: Intracardiac Catheter Ablation — Both arms will receive intracardiac catheter ablation procedures as described.

SUMMARY:
RABLAP-AF will compare pulmonary vein isolation (PVI) in combination with posterior wall isolation (PWI) for patients with persistent atrial fibrillation (AF).

DETAILED DESCRIPTION:
Ablation for AF has a high success rate for patients with paroxysmal AF, but success rates for persistent AF remain significantly lower. These patients frequently have more advanced disease in their left atrium than those with paroxysmal AF.

A common practice is to perform left atrial PWI in addition to PVI in order to reduce AF recurrence. This approach has conflicting evidence behind it and a large scale clinical trial in those with advanced disease is required. The investigators hope to fill this gap with RABLAP-AF.

The investigators will randomise patients with advanced atrial disease 1:1 to PVI+PWI or PVI alone. All patients will receive implantable loop recorders two months prior to the ablation procedure in order to accurately assess the effect of PWI and compare arrhythmia burden before and after ablation.

ELIGIBILITY:
Inclusion criteria:

* Age 18 to 80 (inclusive)
* Patients with symptomatic advanced persistent AF, defined as:
* AF which does not spontaneously terminate and requires medical intervention (antiarrhythmics or DCCV) to terminate, AND
* Recurs following cardioversion, AND
* Is associated with evidence of left atrial cardiopathy, defined as at least mild left atrial enlargement on imaging (echo, CT or MRI) as defined by standard values (for example British Society of Echocardiography or European equivalent) - in the event of uncertainty, Principal Investigator discretion is allowed.

Exclusion Criteria

* Any previous catheter (or surgical) ablation for AF (previous ablation for atrial flutter or focal atrial tachycardias are allowable)
* An indwelling atrial septal defect occluder device or anatomical structure that pre-vents free access to the left atrium
* Severe left ventricular systolic dysfunction (ejection fraction less than 35%)
* Recent stroke/transient ischaemic attack within 3 months
* Inability, unwillingness or absolute contraindication to taking an oral anticoagulant medication
* Severe kidney function impairment (eGFR less than 30ml/min/1.73m2)
* Morbid obesity with a body mass index ≥40
* Extreme frailty (a score of 7,8 or 9 on the Rockwood Clinical Frailty Scale)
* Severe valvular heart disease of any kind as assessed by the investigator, with or without a prosthetic valve in place
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Time to first day with ATA burden of 12 hours or greater | From 3 months post ablation to 12 months
  Time to day with atrial tachyarrhythmia burden lasting 12 hours or greater, following a 3 month blanking period post-ablation

SECONDARY OUTCOMES:
Time to first day with ATA burden of 24 hours | From 3 months post ablation to 12 months
  Time to first day with atrial tachyarrhythmia burden of 24 hours, following a 3 month blanking period post-ablation
Time to first day with ATA burden of 60 minutes or greater | From 3 months post ablation to 12 months
  Time to first day with atrial tachyarrhythmia burden of 60 minutes or greater, following a 3 month blanking period post-ablation
Number of patients with >= 75% reduction in cumulative burden of AF between pre-ablation and months 3-12 | 12 months
  AF burden (assessed by loop recorder) will be analysed in the 2 months pre-ablation and compared with the 9 months post-blanking period. This outcome will assess the number of patients who achieve greater than or equal to 75% reduction.
Reduction in burden of AF between pre-ablation and months 3-12 | 12 months
  AF burden (assessed by loop recorder) will be analysed in the 2 months pre-ablation and compared with the 9 months post-blanking period. This outcome will assess the average % reduction in AF burden between these time periods.
Difference in AFEQT questionnaire between baseline and month 12 | 12 months
  Differences in quality of life indicators as measured by the "AF Effect on QualiTy of life survey" (AFEQT) between baseline and 12 month follow-up
Difference in EQ5D questionnaire between baseline and month 12 | 12 months
  Differences in quality of life indicators as measured by the "EuroQol 5 Dimension survey" (EQ5D) questionnaire between baseline and 12 month follow-up
Difference in VAS between baseline and month 12 | 12 months
  Differences in quality of life indicators as measured by "Visual Analogue Scale" (VAS) between baseline and 12 month follow-up
Use of antiarrhythmic drugs from month 3 onwards | From 3 months post ablation to 12 months
  Number of patients requiring antiarrhythmic drugs following the 3 month blanking period.
Use of direct current cardioversion or repeat ablation | From 3 months post ablation to 12 months
  Number of patients requiring cardioversion or repeat ablation

OTHER OUTCOMES:
Safety Outcome: Number of patients with procedural complications (<2 months post procedure) | Within 2 months of protocol-required invasive procedures
  Number of patients suffering a procedure-related complication within 2 months of an invasive procedure as defined in the study protocol
Safety Outcome: Number of patients undergoing planned and unplanned cardiovascular-related hospitalisations | 12 months
  Number of patients who are hospitalised (planned or unplanned) for cardiovascular reasons

CONTACTS AND LOCATIONS:
Overall Officials: Dhiraj Gupta, MD, Principal Investigator — Liverpool Heart & Chest Hospital
Locations (1):
- Liverpool Heart & Chest Hospital, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No